CLINICAL TRIAL: NCT06977581
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Parallel-group, Dose-Ranging Study to Investigate the Efficacy and Safety of PF-07275315 in Adult Participants With Inadequately Controlled Moderate-to-Severe Asthma
Brief Title: A Study to Learn About the Study Medicine Called PF-07275315 in People With Moderate-To-Severe Asthma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C4531029; 2024-517866-40-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2025-04-25; First posted 2025-05-18 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Asthma
Keywords: Pulmonary; Wheezing; Respiratory hypersensitivity; Airway Inflammation; Airway Obstruction; Dyspnea; Lung Diseases; Respiratory Tract Diseases; Asthma
MeSH Terms: conditions — Asthma; Respiratory Sounds; Respiratory Hypersensitivity; Airway Obstruction; Dyspnea; Lung Diseases; Respiratory Tract Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment Arm A (Experimental): PF-07275315
  Interventions: Drug: PF-07275315
- Treatment Arm B (Experimental): PF-07275315
  Interventions: Drug: PF-07275315
- Treatment Arm C (Experimental): PF-07275315
  Interventions: Drug: PF-07275315
- Treatment Arm D (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: PF-07275315 — subcutaneous injection
  Arms: Treatment Arm A; Treatment Arm B; Treatment Arm C
Other: Placebo — subcutaneous injection
  Arms: Treatment Arm D

SUMMARY:
The purpose of this clinical trial is to learn about the safety and effects of the study medicine (called PF-07275315) for the potential treatment of moderate-to-severe asthma. Asthma is a condition that makes it challenging to breathe, which negatively impacts the quality of life and functioning of people who are affected.

This study is seeking participants who:

* Are 18 to 70 years old
* Have had moderate-to-severe asthma for at least 12 months that is not well controlled
* Have been taking their regular maintenance treatment(s) for asthma over the last 12 months

All participants will receive PF-07275315 or a placebo. A placebo does not have any medicine in it but looks just like the medicine being studied.

PF-07275315 or placebo will be given as multiple shots in the clinic over the course of 12 weeks. We will compare the experiences of people receiving PF-07275315 to those of the people who do not. This will help us determine if PF-07275315 is safe and effective.

Participants will be involved in this study for about 9.5 months. During this time, they will have 10 visits at the study clinic.

ELIGIBILITY:
Inclusion Criteria:

Must meet the following asthma criteria:

1. History of persistent, moderate-to-severe asthma for at least 12 months prior to screening.
2. Must have experienced at least 1 asthma exacerbation requiring treatment with systemic steroids (oral or parenteral) for 3 days or more within 12 months of the screening visit.
3. Pre-bronchodilator FEV1 of ≥30% to <80% of predicted normal values during screening period.
4. Positive bronchodilator responsiveness as evidenced by increase in FEV1 of at least 12% and 200 mL for spirometry conducted during screening period.
5. Maintenance (controller) treatment that minimally includes a medium to high dose ICS - LABA combination consistent with GINA Step 4/5 (either Track 1 or Track 2) for 12 months prior to the screening visit and at a stable dose for at least 3 months prior to the screening visit.
6. ACQ-5 score of ≥1.5 at screening visit and prior to randomization.

   Other Inclusion Criteria:
7. Body mass index between 18 40 kg/m2 at screening.

Exclusion Criteria:

Medical Conditions:

1. Any medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
2. Evidence of lung disease(s) other than asthma, either clinical evidence, spirometry, or imaging (Chest X-ray, CT, MRI) within 12 months of the screening visit, as per local standard of care, including but not limited to: Chronic obstructive pulmonary disease, Other emphysematous lung disease such as alpha-1 antitrypsin disease, Cystic fibrosis, Emphysema, Idiopathic pulmonary fibrosis, Churg-Strauss syndrome, Allergic bronchopulmonary aspergillosis, Sarcoidosis
3. Diagnosed with any of the following acute or chronic infections or infection history:

   * Active helminth or parasitic infection requiring treatment within 2 weeks prior to screening;
   * Infection requiring hospitalization or systemic (parenteral) antimicrobial therapy within 60 days prior to Day 1;
   * Any infection judged to be an opportunistic infection or clinically significant by the investigator, within 6 months prior to Day 1.

   Prior/Concomitant Therapy:
4. Prior or current use of any prohibited concomitant medication(s) or unwillingness or inability to use a required concomitant medication(s).
5. Prior or concurrent treatment with either approved or experimental biologic treatment (such as inhibitors of IL-4Rα, TSLP, IL-5, or IgE) or targeted synthetic drugs (such as JAK inhibitors) for the treatment of asthma or other type 2 inflammatory diseases, including but not limited to: AD, EoE, CRS.
6. Treatment with any dose level of systemic (oral or injectable) corticosteroids within 28 days of the screening visit through the end of study (except to treat an acute exacerbation).
7. Prior (within 12 weeks prior to screening) or planned concomitant treatment with immunoglobulin supplementation (eg, IV Ig or SC Ig).
8. History of anaphylaxis to antibody therapeutic or to PF-07275315 or to the excipients of the formulated drug products.
9. Bronchial thermoplasty within the previous 24 months.

   Prior/Concurrent Clinical Study Experience:
10. Administration of an investigational drug product within 30 days or 5 half lives preceding the screening visit (whichever is longer). Participation in studies of other investigational products (drug or vaccine) at any time during participation in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2027-03-28 (Estimated); Study Completion 2027-08-15 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in pre-bronchodilator Forced Expiratory Volume in 1 Second (FEV1) at Week 12 | Week 12
  FEV1 is the maximal volume of air exhaled in the first second of a forced expiration from a position of full inspiration. FEV1 is obtained from spirometry.
Treatment-Emergent Adverse Events (AEs), Serious AEs (SAEs), and AEs/SAEs leading to treatment discontinuation | Baseline through Week 32
  Incidence of treatment-emergent AEs, treatment-emergent SAEs, and treatment-emergent AEs/SAEs leading to treatment discontinuation
Clinically significant, treatment-related laboratory abnormalities | Baseline through Week 32
  Incidence of clinically significant changes in laboratory tests
Clinically significant, treatment-related abnormalities in vital signs | Baseline through Week 32
  Incidence of clinically significant changes in vital signs
Clinically significant, treatment-related electrocardiogram (ECG) abnormalities | Baseline through Week 32
  Incidence of clinically significant changes in ECG

SECONDARY OUTCOMES:
Change from baseline in pre-bronchodilator Percent (%) Predicted FEV1 at Week 12 | Week 12
Change from baseline in pre-bronchodilator FEV1 at all time points | Baseline through Week 32
Change from baseline in pre-bronchodilator % Predicted FEV1 at all time points | Baseline through Week 32
Change from baseline in pre-bronchodilator Forced Vital Capacity (FVC) at all time points | Baseline through Week 32
Change from baseline in pre-bronchodilator % Predicted FVC at all time points | Baseline through Week 32
Change from baseline in pre-bronchodilator FEV1/FVC Ratio at all time points | Baseline through Week 32
Change from baseline in post-bronchodilator FEV1 at all time points | Baseline through Week 32
Change from baseline in post-bronchodilator % Predicted FEV1 at all time points | Baseline through Week 32
Change from baseline in post-bronchodilator FVC at all time points | Baseline through Week 32
Change from baseline in post-bronchodilator % Predicted FVC at all time points | Baseline through Week 32
Change from baseline in post-bronchodilator FEV1/FVC Ratio at all time points | Baseline through Week 32
Change from baseline in FEV1 as a % of pre-bronchodilator result | Baseline through Week 32
Change from baseline in pre-bronchodilator FEV1 at Week 12 | Week 12
Change from baseline in Asthma Control Questionnaire-5 (ACQ-5) total score at Week 12 | Week 12
Change from baseline in Asthma Quality of Life Questionnaire (AQLQ) global score at Week 12 | Week 12
Change from baseline in pre-bronchodilator FEV1 at Week 12 in participants with Fractional Concentration of Exhaled Nitric Oxide (FeNO) ≥25 ppb and <25 ppb | Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (16):
- United States (11):
  - Velocity Clinical Research, Mobile, Mobile, Alabama
  - Antelope Valley Clinical Trials, Lancaster, California
  - Allergy and Asthma Associates of Santa Clara Valley Research Center, San Jose, California
  - Allergy & Asthma Clinical Research, Walnut Creek, California
  - Circuit Clinical / Impact Medical Allergy, Asthma & Immunology, Riverdale, New Jersey
  - OK Clinical Research, Edmond, Oklahoma
  - Allergy, Asthma and Clinical Research, Oklahoma City, Oklahoma
  - Clinical Research of Rock Hill, Rock Hill, South Carolina
  - Premier Research Center, LLC, Hendersonville, Tennessee
  - Alina Clinical Trials, LLC., Dallas, Texas
  - Greater Heights & Memorial Pulmonary and Sleep, Houston, Texas
- China (2):
  - The Third Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
- Japan (3):
  - National Hospital Organization Osaka Minami Medical Center, Kawachi-Nagano, Osaka
  - NHO Kinki Chuo Chest Medical Center, Sakai, Osaka
  - Fukuwa Clinic, Chuo-ku, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4531029